CLINICAL TRIAL: NCT03395665
Title: Estradiol, Progesterone and Endometrial Thickness in Frozen Euploid Embryo Transfer
Status: Completed | Type: Observational
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Buenaventura Coroleu, Head of Reproductive Medicine Service, Fundacion Dexeus
Other Study IDs: SMD-2018-01
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Infertility; Preimplantation Genetic Diagnosis/Screening; Miscarriage
MeSH Terms: conditions — Infertility; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Estradiol level — Estradiol level measured at previous day of embryo transfer procedure
Other: Progesterone level — Progesterone level measured at previous day of embryo transfer procedure
Other: Endometrial thickness — Endometrial thickness measured at previous day of embryo transfer procedure

SUMMARY:
The development and improvement in Preimplantation genetic diagnosis/screening (PGS) in association with the efficacy and security of vitrification and trophectoderm biopsy, more efficient stimulation schemes and laboratory improvements in culture and embryo selection have contributed to high success of the assisted reproductive technologies(ART). Transferring an euploid embryo avoids one of the main reasons of miscarriage and implantation failure ( Rubio et al, 22016) and overcomes one of the most important confounding factors. Usually, the transfer of euploid embryos is performed under standard hormone replacement therapy (HRT) and are referred to as FET-PGS cycles( Frozen embryo transfer). The study of FET-PGS cycles with the transfer of a single euploid blastocyst is the best model for evaluation of the impact of the endometrial preparation . Among factors influencing FET outcomes, patient's age, endometrial preparation, endometrium thickness, endometrial pattern, number and quality of embryos transferred , difficulty at ET, recently P4 have received more attention .

The importance of Progesterone (P4) in embryo implantation has been widely studied. P4 plays an important role in endometrial gland formation, embryonic implantation and pregnancy maintenance, both in natural and artificial cycles.

ELIGIBILITY:
Inclusion Criteria:

* Frozen embryo transfer (FET) of at least one single euploid embryo.
* Estradiol > 75pg/ml.
* Progesterone > 4 ng/ml.
* Endometrial thickness between 6 mm and 18 mm.

Exclusion Criteria:

* Patients with FET of no diagnostic or mosaic embryos, or known uterine abnormality were excluded.
* Natura cycle protocol.

Ages: 18 Years to 43 Years | Sex: Female
Age Groups: Adult
Study Population: Women who underwent blastocyst trophectoderm biopsy and PGS and frozen-thawed embryo transfers(PGS-FET) performed after the In Vitro Fertilization (IVF) .
  PGS was implemented as 46-chromosome screening, using array comparative genomic hybridization (aCGH) from Day 5 trophectoderm biopsy. Whole-genome amplification, processing and analyses were performed using the kits, software and protocols for array Comparative Genomic Hybridisation (aCGH) analysis provided by the manufacturer (SurePlex® DNA Amplification System, 24Sure® Microarray Pack, Bluefuse®, Illlumina®).
Sampling Method: Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Live birth rate | Ten months after transfer procedure
Miscarriage rate | Any pregnancy loss before week 20
  Miscarriage was defined as a loss following a positive pregnancy test and/or detectable Gestational sac
Pregnancy rate | 6 weeks after transfer procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics, Gynaecology and Reproduction Instituto Universitario Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.dexeus.com